CLINICAL TRIAL: NCT03115749
Title: Characterization of Mesenchymal Stem Cells From the Colon and Small Intestine of Patients With Inflammatory Bowel Disease - The COSMIC Study
Brief Title: Intestinal Mesenchymal Stem Stells and Inflammatory Bowel Diseases
Acronym: COSMIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period and recruitment difficulties
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9755
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease; ulcerative colitis; mesenchymal stem cells; intestinal inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crohn's disease patient group (Other): Intestinal biopsies during colonoscopy or biopsies taken on surgical specimen after intestinal resection
  Interventions: Other: Intestinal biopsies during colonoscopy; Other: Biopsies taken on surgical specimen
- Ulcerative colitis patient group (Other): Intestinal biopsies during colonoscopy or biopsies taken on surgical specimen after intestinal resection
  Interventions: Other: Intestinal biopsies during colonoscopy; Other: Biopsies taken on surgical specimen
- Control group (Other): Intestinal biopsies during colonoscopy or biopsies taken on surgical specimen after intestinal resection
  Interventions: Other: Intestinal biopsies during colonoscopy; Other: Biopsies taken on surgical specimen

INTERVENTIONS:
Other: Intestinal biopsies during colonoscopy — Intestinal biopsies during colonoscopy
Other: Biopsies taken on surgical specimen — biopsies taken on surgical specimen after intestinal resection

SUMMARY:
The exact origin of inflammatory bowel disease (IBD) is still unknown. The current hypothesis is that IBD is secondary to an abnormal intestinal immun response directed to all or part of the intestinal flora in genetically predisposed individuals. Several experimental studies have demonstrated the ability of mesenchymal stem cells (MSCs) from bone marrow or adipose tissue origin to control intestinal inflammation in animal models. However, to date, there are no data regarding the functions of resident MSCs in the colon and small intestine of IBD patients. We hypothesize that dysfunction of resident intestinal MSCs contributes to the disruption of intestinal homeostasis in patients with IBD causing the development of intestinal inflammation. The aim of this research project is to identify, describe and characterize at the molecular and functional level MSCs of the colon and small intestine of patients with Crohn's disease and ulcerative colitis and to compare them with a control population.

DETAILED DESCRIPTION:
Primary and secondary objectives:

Main Objective: Characterize morphologically, molecularly and functionally the MSCs of colon and small intestine of patients with IBD and compared to MSCs of colon and small intestine of control patients.

Secondary objectives: To study the reaction of colon and small intestine MHC in patients with IBD following stimulation with bacterial compounds.

Methodology:

Clinical study exploratory translational physiopathological. Two groups of patients with Crohn's disease and ulcerative colitis who require colonoscopy or surgery for intestinal resection will be included. These two groups will be compared to a control group consisting of patients requiring colonoscopy for screening or intestinal resection for colorectal cancer or diverticulum.

Intestinal sampling by biopsy during the colonoscopy or with surgical specimen during the surgery will be performed to isolate the MSCs.

The outcome measures will be a qualitative and quantitative analysis of MSCs by immunohistochemistry, immunofluorescence, cell proliferation and differentiation, production of pro- and anti-inflammatory cytokines in the basal state and after bacterial stimulation.

Total of 60 patients (20 in groups, 15 with colonoscopy and 5 with surgical specimens).

ELIGIBILITY:
Inclusion criteria:

* For IBD patients :

  * Age between 18 and 75 year old
  * Diagnosis of Crohn's disease or ulcertaive colitis according to internationla guidelines
  * Endoscopically active disease
  * Indication for colonoscopy or intestinal resection according to standard of care
  * Written inform consent
* For control patients :

  * Age between 18 and 75 year old
  * Indication for screening colonoscopy for irritable bowel syndrome, diverticulum or colorectal cancer surveillance according to standard of care
  * Indication for intestinal resection for diverticulum or colorectal cancer according to standard of care
  * Written inform consent

Exclusion criteria:

* For IBD patients :

  * Active intestinal infection
  * Confirmed intestinal parasitosis
  * Intestinal stoma
* For control patients :

  * Active intestinal infection
  * Confirmed intestinal parasitosis
  * Intestinal inflammation at colonoscopy
  * Chronic intestinal inflammation on biopsies
  * Absence of healthy tissue on surgical specimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Proliferation and differentiation of intestinal MSCs in IBD patients. | 1 month
  Proliferation and differentiation of intestinal MSCs in IBD patients.

SECONDARY OUTCOMES:
Comparison of MSCs between IBD patients and control patients | 1 month
  Comparison of MSCs between IBD patients and control patients using mmunohistochemistry, immunofluorescence, quantification of pro- and anti-inflammatory cytokines production.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pineton de Chambrun, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hopital St Eloi, Montpellier, France

IPD SHARING:
Plan to Share IPD: No